CLINICAL TRIAL: NCT01990872
Title: Randomized Controlled Trial to Explore the Inter-relationship Between Vitamin D Requirements and Calcium Intake
Brief Title: Inter-relationship Between Vitamin D Requirements and Calcium Intake in Older Adults
Acronym: VitD-Ca
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Kevin D. Cashman, Professor of Food and Health, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PR-IC-1111-10005
Record Dates: First submitted 2013-11-08; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D status; 25-hydroxyvitamin D; Vitamin D3; RCT; Calcium intake; Dietary requirement
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo in high calcium group (Placebo Comparator): Placebo + habitual dietary calcium intake (>1000 mg/d)
  Interventions: Dietary Supplement: Placebo
- Vitamin D3 in low/moderate calcium group (Active Comparator): Vitamin D3 (20 microgram/day) + habitual calcium intake <700 mg/d
  Interventions: Dietary Supplement: Vitamin D3 (20 micrograms/day)
- Placebo in low/moderate calcium group (Placebo Comparator): Placebo + habitual calcium intake <700 mg/d
  Interventions: Dietary Supplement: Placebo
- Vitamin D3 in high calcium group (Active Comparator): Vitamin D3 (20 microgram/day) + habitual calcium intake (>1000 mg/d)
  Interventions: Dietary Supplement: Vitamin D3 (20 micrograms/day)

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (20 micrograms/day) — Vitamin D3 (20 micrograms/day)
  Arms: Vitamin D3 in high calcium group; Vitamin D3 in low/moderate calcium group
Dietary Supplement: Placebo — Placebo (0 micrograms vitamin D3/day)
  Arms: Placebo in high calcium group; Placebo in low/moderate calcium group

SUMMARY:
This winter-based placebo-controlled, single-dose vitamin D randomized controlled trial (RCT) aims to examine the impact of various levels of habitual calcium intake on dietary vitamin D requirements in older adults stratified by calcium intake. This will provide new data on the impact of different levels of calcium intake, ranging from low/moderate to high, on winter serum 25(OH)D levels, and their utilization and catabolism in adults.

DETAILED DESCRIPTION:
The aim of this study is to perform a randomised controlled vitamin D3 intervention study in apparently healthy, free-living adults (aged 50+ y) to investigate whether different levels of habitual calcium intake, ranging from low-moderate to high, influence serum 25(OH)D concentrations and indices of vitamin D activation and catabolism during winter, when vitamin D intake is adequate versus inadequate.

This research will provide new data and scientific understanding in relation to the impact of different levels of dietary calcium intake on vitamin D requirements in the older adult population. As such, this new data will inform dietary reference values for vitamin D.

ELIGIBILITY:
Inclusion Criteria:

Consenting white men and women aged ≥ 50 y

Exclusion Criteria:

* Unwilling to discontinue consumption of vitamin D-containing supplements 4 wks before the initiation of the study and throughout the study.
* Planning to take a winter vacation (during the course of the 15-wk intervention) to a location at which either the altitude or the latitude was predicted to result in significant cutaneous vitamin D synthesis from solar radiation (e.g., a winter sun coastal resort or a mountain ski resort)
* Use of tanning facilities of any type.
* Pregnancy or planning to become pregnant during the study
* A severe medical illness,
* hypercalcaemia,
* Known intestinal malabsorption syndrome,
* Excessive alcohol use,
* Taking medications known to interfere with vitamin D metabolism

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Response of serum 25(OH)D concentration over winter in subjects stratified by calcium intake | 0, 8, 15 weeks

SECONDARY OUTCOMES:
Serum albumin-adjusted calcium | 0, 8, 15 weeks
serum parathyroid hormone | 0, 8, 15 weeks
Serum 24,25(OH)2D | 0 and 15 weeks
Serum 1,25(OH)2D | 0 and 15 weeks
Serum free 25(OH)D | 0 and 15 weeks
Serum vitamin D binding protein | 0 and 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D Cashman, BSc. PhD, Principal Investigator — University College Cork
Locations (1):
- Human Dietary Studies Facility, School of Food and Nutritional Sciences, University College Cork, Cork, Ireland, Cork, Ireland

REFERENCES:
- [Derived] Cashman KD, Kinsella M, Walton J, Flynn A, Hayes A, Lucey AJ, Seamans KM, Kiely M. The 3 epimer of 25-hydroxycholecalciferol is present in the circulation of the majority of adults in a nationally representative sample and has endogenous origins. J Nutr. 2014 Jul;144(7):1050-7. doi: 10.3945/jn.114.192419. Epub 2014 May 14. PMID 24828024
- [Derived] Cashman KD, Hayes A, O'Donovan SM, Zhang JY, Kinsella M, Galvin K, Kiely M, Seamans KM. Dietary calcium does not interact with vitamin D(3) in terms of determining the response and catabolism of serum 25-hydroxyvitamin D during winter in older adults. Am J Clin Nutr. 2014 Jun;99(6):1414-23. doi: 10.3945/ajcn.113.080358. Epub 2014 Apr 2. PMID 24695896